CLINICAL TRIAL: NCT07160010
Title: Clinical Validation of Sophia Genetics Assays on MGI Sequencing Platform
Brief Title: Clinical Validation of Sophia Genetics Assay
Acronym: COSMOS
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7180
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Breast Cancer; Lynch Syndrome; Intestinal Polyposis
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis; Intestinal Polyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sophia Herditary Cancer Solution — To compare the performance of MGI's DNBSEQ-G400 sequencing instrument with the gold standard Illumina instruments (MiSeq and NextSeq 550) using the same capture DNA libraries constructed with Sophia Genetics assays.
  Other Names: Sophia Exome Clinical Solutions v3

SUMMARY:
Next-generation sequencing (NGS) technologies have revolutionized the field of genomics, enabling rapid and cost-effective analysis of DNA and RNA . Among NGS methods, Illumina sequencing is the most widely used, due to its high-throughput and parallel sequencing capabilities. Nanopore sequencing, passes DNA through a nanopore, and the sequence is identified based on changes in electrical current. MGI's sequencing platforms use combinatorial probe-anchor synthesis technology to achieve high-throughput sequencing. These diverse NGS techniques have broad applications, including genome sequencing, metagenomics, and epigenetics, offering powerful tools for exploring genetic information.The main distinction between MGI and Illumina platforms lies in their methods for constructing and amplifying sequencing libraries. DNBSEQ™ utilizes circular single-stranded libraries with a central adapter, which are amplified by a rolling circle replication system to produce DNA nanoballs (DNBs). Each DNB then binds to a flowcell well via ionic bonds. Illumina technology employs linear double-stranded libraries with adapters at both ends, which are hybridized and amplified in clusters using bridge PCR. Both platforms use ordered flowcells and sequencing-by-synthesis methods. Thanks to its linear DNB amplification approach, where each replica is generated from the same original template, DNBSEQ™ technology eliminates detectable clonal amplification errors (specific to PCR) and index hopping, while also producing a very low rate of duplicated sequences. The MGI sequencer can accommodate two flowcells in parallel, each divided into four independent lanes. It is compatible only with MGI library preparation kits, while analysis pipelines developed for Illumina data are also compatible with MGI data.This study aims to compare the performance of MGI's DNBSEQ-G400 sequencing instrument with the gold-standard Illumina instruments (MiSeq and NextSeq 550) using the same DNA capture libraries constructed with Sophia Genetics assays. The goal is to assess whether MGI's platform is comparable to Illumina in profiling patients with solutions commercialized by Sophia Genetics.

ELIGIBILITY:
Inclusion Criteria:

* Samples from patients with hereditary breast and ovarian cancer (HBOC), Lynch syndromes, and intestinal polyposis that will undergo genetic testing with commercial solutions provided by Sophia Genetics and sequenced on Illumina;
* Samples from patients with rare and hereditary disorders that have been profiled with commercial solutions provided by Sophia Genetics and sequenced on Illumina;
* Samples of patients for whom a report of the results is available;
* Samples of patients who have previously consented and are aware if their genomic results.

Exclusion Criteria:

* patients for whom blood, DNA or tissue samples are not available for analysis;
* samples that do not pass the quality check, set as DNA concentration, DNA integrity, library concentration and quality;
* samples for which consent for future analysis has not be given.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve samples from patients with hereditary breast and ovarian cancer (HBOC), Lynch syndrome, and intestinal polyposis, who will undergo genetic testing using commercial solutions from Sophia Genetics, sequenced on Illumina platforms. It will also include samples from patients with rare and hereditary disorders, profiled using Sophia Genetics' commercial solutions and sequenced on Illumina platforms. Additionally, samples from patients with available genetic test reports will be included, as well as samples from patients who have previously consented and are aware of their genomic results.
Sampling Method: Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparation between sequencing platforms | 12 months
  To assess whether MGI's platform is superimposable with Illumina in profiling patients with solutions commercialized by Sophia Genetics.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Minucci, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS